CLINICAL TRIAL: NCT00181155
Title: Effects of Xanthine Oxidase Inhibition on Mechano-Energetic Coupling in Heart Failure
Brief Title: Intravenous Allopurinol in Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert G. Weiss, Professor of Medicine and Radiology, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB: 04-10-12-06; 5R01HL061912-14 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Congestive Heart Failure
Keywords: metabolism; congestive heart failure; allopurinol; Adenosine triphosphate (ATP)
MeSH Terms: conditions — Heart Failure | interventions — Allopurinol; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Experimental): One time intravenous administration of Allopurinol 300 mg infused over approximately 20 minutes.
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): One time intravenous administration of 50 ml dose of 5% dextrose infused over approximately 20 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allopurinol — intravenous infusion of allopurinol (300mg)
  Other Names: Aloprim
  Arms: Allopurinol
Drug: Placebo — intravenous infusion of 50 ml dose of 5% dextrose
  Other Names: 5% Dextrose
  Arms: Placebo

SUMMARY:
This study tests the hypothesis that allopurinol, a xanthine oxidase inhibitor, improves heart metabolism in patients with heart failure.

DETAILED DESCRIPTION:
Xanthine oxidase have been reported to improve mechano-energetic coupling in failing hearts. The investigators developed a means to directly measure creatine kinase flux, the major energy reserve of the heart, in the human heart exploiting new magnetic resonance technologies.

The investigators propose to study 10 healthy subjects and up to 25 with heart failure (dilated cardiomyopathy) before and after a single 300mg IV infusion of allopurinol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* The patient is willing and able to provide informed consent
* Clinical diagnosis of chronic heart failure
* Ejection fraction (EF) < 40% by echocardiography, nuclear multigated acquisition (MUGA) or cath ventriculography
* No significant coronary disease at cardiac catheterization
* New York Heart Association (NYHA) Class I-IV symptoms
* Clinical stabilization for two weeks if following recent congestive heart failure (CHF) decompensation.

Exclusion Criteria:

* Metallic implant prohibiting magnetic resonance (MR) evaluation
* Inability to lie flat for MR study
* Administration of additional investigational drugs
* Calculated creatinine clearance < 50 mL/min
* Allergy to allopurinol
* Current gout flare
* Currently taking oral allopurinol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Weiss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hirsch GA, Bottomley PA, Gerstenblith G, Weiss RG. Allopurinol acutely increases adenosine triphospate energy delivery in failing human hearts. J Am Coll Cardiol. 2012 Feb 28;59(9):802-8. doi: 10.1016/j.jacc.2011.10.895. PMID 22361399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Non-Ischemic Cardiomyopathy were recruited as approved by the Johns Hopkins Institutional Review Board for Human Investigation.
Pre-assignment Details: The study drug allocation was randomized in a 4:1 fashion by the research pharmacy. Participants were randomized to Placebo only for the purposes of blinding; Adverse Events were collected for the Placebo arm.
Groups:
- Allopurinol; Placebo: Each participant underwent magnetic resonance spectroscopy before and following infusion of either allopurinol 300mg or placebo.
Period: Overall Study
Arm/Group | Allopurinol | Placebo
Started | 15 | 3
Completed | 13 | 3
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intravenous Allopurinol: We randomized patients with nonischemic cardiomyopathy in a double-blind fashion to allopurinol (300 mg intravenously) or placebo infusion, 4-to-1, the latter for purposes of blinding only. The myocardial concentrations of ATP and creatine phosphate (PCr) and the rate of adenosine triphosphate (ATP) synthesis through CK (CK flux) were determined by 31-Phosphorus (31P) magnetic resonance spectroscopy.
Arm/Group | Intravenous Allopurinol
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Creatine Kinase (CK) Flux Pre Intravenous Allopurinol Infusion
Description: Magnetic resonance spectroscopy (MRS) Measurement of Myocardial CK Flux Pre Intravenous Allopurinol Infusion
Time Frame: Onset of imaging acquisition.
Population: Data were analyzed for all participants who completed the MRS per protocol.
Measure: Mean (Standard Deviation); unit: umol/g/sec
Groups:
- Baseline: Each participant underwent baseline MRS imaging prior to infusion of Aloprim 300 mg in 50 cc of 5% Dextrose.
Arm/Group | Baseline
Number analyzed (Participants) | 13
umol/g/sec | 2.07 (1.27)

2. Secondary Outcome: Cardiac PCr/ATP Pre Intravenous Infusion
Description: The mean ratio of creatine phosphate (PCr) to ATP in the heart. This measure, as a ratio, is unitless.
Time Frame: Onset of image acquisition.
Population: Data were analyzed for all participants who completed the MRS per protocol.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Baseline
Number analyzed (Participants) | 13
ratio | 1.58 (0.41)

3. Primary Outcome: Myocardial CK Flux Post Intravenous Allopurinol Infusion.
Description: The mean rate of adenosine triphosphate (ATP) flux through the creatine kinase reaction in the heart.
Time Frame: acute (within 15 minutes of single infusion)
Population: Data were analyzed for all participants who completed the MRS per protocol.
Measure: Mean (Standard Deviation); unit: umol/g/sec
Groups:
- Intravenous Allopurinol: Infused Aloprim 300 mg in 50cc 5% dextrose. Post MRS data acquired on each subject.
Arm/Group | Intravenous Allopurinol
Number analyzed (Participants) | 13
umol/g/sec | 2.87 (1.82)
Statistical Analysis 1: Comparison: Intravenous Allopurinol; Test type: Superiority or Other; p < 0.007, Two-sided paired t tests — vs. baseline

4. Secondary Outcome: Cardiac PCr/ATP Post Intravenous Infusion
Description: The mean ratio of creatine phosphate (PCr) to ATP in the heart. This measure, as a ratio, is unitless.
Time Frame: acute (within 15 minutes of single infusion)
Population: Data were analyzed for all participants who completed the MRS per protocol.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Intravenous Allopurinol: Infused Aloprim 300 mg in 50cc of 5% dextrose. Post infusion MRS data acquired on each subject.
Arm/Group | Intravenous Allopurinol
Number analyzed (Participants) | 13
ratio | 1.75 (0.59)
Statistical Analysis 1: Comparison: Intravenous Allopurinol; Test type: Superiority or Other; p < 0.02, Two-sided paired t tests — vs. baseline

ADVERSE EVENTS:
Groups:
- Arm 1 - Intravenous Allopurinol: Each participant received pre and post MRS images following infusion of 50 cc of Aloprim 300mg in 5% Dextrose.
- Arm 2 - Placebo: Each participant received pre and post MRS images following infusion of 50 cc of 5% Dextrose (equivalent volume to active treatment arm).
Arm/Group | Arm 1 - Intravenous Allopurinol | Arm 2 - Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/3
Other Adverse Events (participants affected / at risk) | 0/13 | 0/3

LIMITATIONS AND CAVEATS:
The limitations of the current study include the small placebo group sample size and the etiologic heterogeneity of the nonischemic cardiomyopathy group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No